CLINICAL TRIAL: NCT06723275
Title: Validation of LEOPARD Predictive Models of Delisting in Liver Transplant Candidates: the LEOPARD Longitudinal Multicentre Prospective Validation Cohort 1, with Bio- and Tissue Collection
Brief Title: LEOPARD Prospective Validation Cohort 1
Acronym: LEOPARD PVC1
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Luxembourg (Other); Hospital Universitario La Fe (Other); ECRIN EUROPEAN CLINICAL RESEARCH INFRASTRUCTURE NETWORK (ECRIN) (Unknown); Ophiomics - Precision Medicine (Unknown); EF CLIF (Unknown); INSERM 1149 (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP231778; 2024-A00808-39 (Other: ID-RCB)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Decompensated Liver Cirrhosis; Primary Biliary Cholangitis; Primary Sclerosing Cholangitis; Hepato-cellular Carcinoma
Keywords: Liver transplantation; Predictive models; Liver transplantation candidates; prospective longitudinal study
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For patients of subsets 1 and 2 :
  * Blood - 3 Dry tubes and 2 EDTA 5mL
  * Blood - 2 EDTA, 1 Li heparin, 2 citrate 5mL
  * Blood - 1 Tempus 10mL biobanking for DNA, RNA
  * Urine 1 plastic tube 5mL
  * Urine 1 hemolysis tube 5 mL
  * Ascites fluid 1 Dry tube 5mL
  For patients of subset 3 :
  * Blood - 1 Streck 10mL
  * Blood - 1 EDTA 5mL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subset 1: Decompensated cirrhosis as primary diagnosis, irrespective of liver disease etiology
  Interventions: Other: Standardized assessments and biobanking
- Subset 2: Other chronic end-stage liver diseases requiring LT, listed under MELD offering schemes, including notably but not exclusively cholestatic diseases, primary biliary cholangitis, primary sclerosing cholangitis
  Interventions: Other: Standardized assessments and biobanking
- Subset 3: Hepato-cellular carcinoma as primary diagnosis, whatever the etiology of the underlying liver disease with or without underlying cirrhosis
  Interventions: Other: Standardized assessments, guided tumor biopsy and biobanking

INTERVENTIONS:
Other: Standardized assessments, guided tumor biopsy and biobanking — Standardized assessment of Scores
  * Guided tumor biopsy in patients listed for hepatocellular carcinoma with active tumor at listing in centers not perfoming tumor biopsy on a routine basis
  * Additional blood sampling for biobanking and subsequent analysis of innovative biomarkers and OMICs
  * Urine sampling for biobanking and subsequent analysis of innovative biomarkers
  * Ascite sampling for biobanking and subsequent analysis
  * Tumor sampling for biobanking and subsequent analysis
  * Centralized assay for routine biomarkers
  Groups: Subset 3
Other: Standardized assessments and biobanking — * Standardized assessment of Scores
  * Additional blood sampling for biobanking and subsequent analysis of innovative biomarkers and OMICs
  * Urine sampling for biobanking and subsequent analysis of innovative biomarkers
  * Ascite sampling for biobanking and subsequent analysis
  * Tumor sampling for biobanking and subsequent analysis
  * Centralized assay for routine biomarkers
  Groups: Subset 1; Subset 2

SUMMARY:
Intro:

The present clinical research protocol is part of the LEOPARD European project (Grant n° 101080964 Horizon Europe) which aims to design and validate new predictive models of mortality among liver transplantation (LT) candidates.

MELD based-liver graft allocation systems have become increasingly inaccurate over the last decade to predict mortality/dropout of liver transplantation (LT) candidates on the waitlist (WL). Wide disparities in mortality/dropout on the WL also exist across European countries, ranging from 5 to 30% according to transplantation indications. In this setting, the European Commission- Horizon Europe funded-LEOPARD project intends to design new, 2nd generation, AI-machine learning-based predictive models of delisting in LT candidates, to better serve on time patients with the highest risk of dropout on the WL and to improve equity of access to LT across Europe.

Hypothesis/Objective The scientific justification of the LEOPARD PVC1 is therefore

1. to build an external cohort of LT candidates to test and validate the LEOPARD models, therefore providing robust evidence for adoption of LEOPARD models by Organ Sharing Organizations (OSOs).
2. to collect granular data, bio- and tissues sampes and images to test last-generation OMICs predictors and radiomics, therefore opening the door to design of 3rd generation, precision medicine-based predictive models.

The primary objective of the LEOPARD longitudinal study is to test and validate AI-based 2nd generation LEOPARD predictive models of mortality/drop out on the waitlist in patients with decompensated cirrhosis, or other end-stage chronic liver diseases, and in patients listed for HCC.

Method Multicenter Prospective longitudinal study in up to 630 enrolments (in case of replacing participants after inclusion) to obtain 600 patients meeting selection criteria, in 30 hospitals in 5 European countries including France, Italy, The Netherlands, Belgium and Germany.

ELIGIBILITY:
Inclusion Criteria:

* Adult [age 18;70] patients listed for:

  * decompensated cirrhosis as primary diagnosis, irrespective of liver disease etiology (subset1) OR
  * other end-stage liver diseases requiring LT, listed under MELD offering schemes (subset 2), including notably but not exclusively cholestatic diseases, primary biliary cholangitis, primary sclerosing cholangitis (subset 2) OR
  * HCC as primary diagnosis, whatever the etiology of the underlying liver disease with or without underlying cirrhosis (subset 3). (HCC diagnosed on Barcelona/EASL criteria or histologically proven. HCC meeting or not Milan criteria, as per center practice.)
* Patients registered on national waiting lists under the MELD offering schemes, regardless of extra MELD points are affected or not.
* Patient (or trusted person, family member or close relation, if the patient is unable to express consent) who has been informed and signed the informed consent.
* Patient affiliated with a health insurance scheme (beneficiary or entitled party).

Exclusion Criteria:

* Tumor vascular invasion (portal or hepatic veins) evidenced by imaging on pre transplantation work-up, including PVT stage 1
* Extra-hepatic metastasis of HCC, as assessed by sectional imaging, functional imaging (18 FDG PET CT/MRI) or histologically proven
* Women who are pregnant or nursing
* Patients who are under safeguard of justice or tutorship or curatorship
* Patient on AME (state medical aid)
* Participation in another trial including other studies proposed as part of the European LEOPARD project (cohort associated to WP1 & WP5 ("LEOPARD TVDCS") or being in the exclusion period following previous interventional research involving the human person, if applicable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients consecutively listed for LT for end-stage chronic liver diseases and HCC
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Clinical primary endpoint will be a composite of mortality or drop out for being too sick on transplantation waiting list, since kinetics of dropout differs according to LT indications | 3 months after listing in subsets 1 & 2 ; 12 months after listing in subset 3
  * 3-month mortality/dropout for being too sick after listing in subsets 1 and 2
  * 12-month mortality/dropout for being too sick (tumor progression) after listing in subset 3

SECONDARY OUTCOMES:
Number of participants with 6-month mortality/dropout for being too sick (subsets 1 to 3) | 6 months after listing
  Mortality/Drop out for being too sick (subsets 1 to 3)
Number of participants with 9-month mortality/dropout for too sick in subsets 1, 2 | 9 months after listing
  Mortality/dropout for being too sick
Number of participants with 12-month mortality/dropout for too sick in subset 3 | 12 months after listing
  Mortality/dropout for being too sick
Causes of death/drop-out for being too sick | From date of inclusion until date of death from any cause or date of drop-out for being too sick, whichever came first, assessed up to 12 months
  Causes of death/drop-out
Incidence of delisting for patient's decision or clinical improvement | From date of inclusion until date of delisting for patient's decision or clinical improvement, assessed up to12 months
  Delisting for patient's decision or clinical improvement
Time from listing to death/drop-out | From date of listing until date of death from any cause or date of drop-out for being too sick, whichever came first, assessed up to 12 months
  Duration from listing to death/dropout (days)
Time to transplantation | From date of listing until date of transplantation, assessed up to 12 months
  Duration from listing to transplantation (days)
Number of participants with 1-year post transplant survival in subsets 1-2 | 12 months after liver transplantation
  Survival in subsets 1-2
Number of participants with 9-month HCC recurrence in subset 3 | 9 months after liver transplantation
  HCC recurrence in subset 3
Number of participants with 9-month post transplant survival in subset 3 | 9 months after liver transplantation
  Post transplant survival in subset 3
9-month and 12-month transplant benefit in subsets 3 and 1-2, respectively | 9 months and 12 months after liver transplantation
  Relevant comorbidities

CONTACTS AND LOCATIONS:
Locations (5):
- Department of Gastroenterology and Hepatology Universitair Ziekenhuis Gent, Ghent, Belgium, Belgium
- Hospital Henri Mondor, Department of Hepatology, Créteil, France, France
- Universitätsklinikum Schleswig - Holstein | UKSH · Transplantation Medicine, Kiel, Germany, Germany
- Italian National Transplant Center, Roma, Italy, Italy
- Center for Liver Tumors Leiden of the Leiden University Medical Center (LUMC), Leiden, Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION